CLINICAL TRIAL: NCT04317794
Title: A Multicenter, Observational, Postmarketing Surveillance Study of Spinraza Injection (Nusinersen Sodium) When Used in Routine Medical Practice in Korea
Brief Title: Observational, Postmarketing Surveillance Study of Spinraza Injection (Nusinersen Sodium)
Acronym: STANDARD
Status: Active, not recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 232SM403
Record Dates: First submitted 2020-03-05; First posted 2020-03-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- All Participants: Participants who were prescribed with nusinersen sodium injection in Korea according to local marketing authorization.
  Interventions: Drug: Nusinersen Sodium Injection

INTERVENTIONS:
Drug: Nusinersen Sodium Injection — Administered as specified in the treatment arm.
  Other Names: BIIB058; ISIS 396443; Spinraza

SUMMARY:
The primary objective is to evaluate the safety of nusinersen sodium injection in the postmarketing setting in Korea. The secondary objective is to evaluate the effectiveness of nusinersen sodium injection in the postmarketing setting in Korea.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently receiving or about to initiate treatment with commercial Spinraza in the postmarketing setting
* Genetic documentation of 5q-linked SMA

Key Exclusion Criteria:

* Hypersensitivity to the active substance or any of the excipients of Spinraza
* Ongoing participation or participation within 6 months or 5 half-lives of the agent (whichever is longer) of enrollment in other interventional clinical trials for the treatment of SMA
* Inability to comply with study requirements

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are receiving or about to initiate treatment with commercial Spinraza in Korea according to the local marketing authorization (including documentation of SMA diagnosis), agree to the collection and use of data as specified in the protocol, and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to End of Treatment (2 Years)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event.

SECONDARY OUTCOMES:
Change from Baseline in Hammersmith Infant Neurological Examination (HINE) Section 2 Scores | Baseline, Day 63 and Approximately Every 4 Months Up to End of Treatment (2 years)
  Section 2 of the HINE is used to assess motor milestones of the participants. It is composed of 8 motor milestone categories: voluntary grasp, ability to kick in supine position, head control, rolling, sitting, crawling, standing, and walking.
Change from Baseline in Hammersmith Functional Motor Scale - Expanded (HFMSE) | Baseline, Day 63 and Approximately Every 4 Months Up to End of Treatment (2 years)
  The HFMSE is a tool used to assess motor function in children with SMA. The original 20 item Hammersmith Functional Motor Scale (HFMS) was expanded to include 13 additional items to improve sensitivity for the higher functioning ambulant population. Participants are asked to complete a specific movement and are then graded on the quality and execution of that movement. Higher scores indicate higher levels of motor ability where 0=unable, 1=performed with some assistance, and 2=unaided. The overall score is the sum of the scores for all activities.
Time to Death | Up to End of Treatment (2 years)
Number of Participants with Ventilatory Support | Up to End of Treatment (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (16):
- South Korea (16):
  - Pusan Natioanl University Hospital, Busan
  - Samsung Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Chonbuk National University Hospital, Jeonju
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea university Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Natioanl University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com
URL: https://vivli.org/